CLINICAL TRIAL: NCT05868993
Title: Optimal Effective Local Anesthetic Volume for Pain Relief Using Brachial Plexus Block Utilizing Continuous Reassessment Method for Arthroscopic Rotator Cuff Shoulder Surgery
Brief Title: Optimal Effective Local Anesthetic Volume for Pain Relief Using Brachial Plexus Block
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benaroya Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB20-018
Record Dates: First submitted 2023-04-27; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-02

CONDITIONS: Post Operative Pain
Keywords: brachial plexus block
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Brachial Plexus Block Group 1 (Experimental): Interscalene
  Interventions: Drug: Dose of 0.5% Ropivacaine
- Brachial Plexus Group 2 (Experimental): Supraclavicular
  Interventions: Drug: Dose of 0.5% Ropivacaine
- Brachial Plexus Group 3 (Experimental): Suprascapular
  Interventions: Drug: Dose of 0.5% Ropivacaine

INTERVENTIONS:
Drug: Dose of 0.5% Ropivacaine — Dose varied by 5mL of 0.5% Ropivacaine

SUMMARY:
Prospective, patient-blinded study utilizing a novel Continuous Reassessment Method that concomitantly considers both block success and block side effects (lung dysfunction) for brachial plexus nerve blocks.

DETAILED DESCRIPTION:
Success or failure of the brachial plexus block for any given volume will be determined by the verbal analogue pain scale score obtained 60 minutes after surgical end time. Volumes will be determined by continuous reassessment method.

ELIGIBILITY:
Inclusion Criteria:

* Surgical candidate for Arthroscopic rotator cuff surgery
* ASA I-III
* BMI<40
* Age >18

Exclusion Criteria:

* Inability to give informed consent
* Inability to complete consent process in English
* allergy to ropivacaine
* neuropathy
* contraindications to peripheral nerve block per ASRA guidelines
* chronic opioid use
* infection at the injection/catheter site
* limb restriction due to medical history
* history of moderate - severe lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Block Success | 60min after surgery
  Block success measured by pain (11-point VAS)
Lung Function | 60 mins after surgery
  Block success as measured by preservation of lung function (Vital Capacity in L)
Block Success | 60 mins after surgery
  Block Success measured by opioid (mcg of fentanyl delivered)

SECONDARY OUTCOMES:
Diaphragm Excursion | 60 minutes after surgery
  Change in Movement of Diaphragm in cm
Vital Capacity | 60 minutes after surgery
  Change in Vital Capacity measured in L
Pulse Oximetry | 60 minutes after surgery
  Change in Pulse Oximetry Value
Side Effects | 60 minutes after surgery
  Rate of Dyspnea, Horner's, Hoarseness

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Mason Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No